CLINICAL TRIAL: NCT03424889
Title: Effect of Xylometazoline Administration During Nasal Flexible Bronchoscopy: A Double Blind, Randomized, Placebo-controlled Trial
Brief Title: Xylometazoline During Nasal Flexible Bronchoscopy
Acronym: VAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Karan Madan, MD DM, Assistant Professor, Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IEC AIIMS/Vasoconstrictor RCT
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Bronchoscopy
Keywords: Bronchoscopy; Lignocaine; Anaesthesia
MeSH Terms: interventions — xylometazoline; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Concealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xylometazoline (Experimental): Patients receiving topical xylometazoline nasally during bronchoscopy
  Interventions: Drug: Xylometazoline
- Saline placebo (Placebo Comparator): Patients receiving topical saline nasally during bronchoscopy
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Xylometazoline — Nasal administration of Xylometazoline
  Arms: Xylometazoline
Drug: Saline — Nasal administration of 0.9% Saline
  Arms: Saline placebo

SUMMARY:
Flexible bronchoscopy is a commonly performed procedure and is usually performed transnasally. The optimal topical anesthesia regimen for bronchoscopy is investigational. Topical Vasoconstrictors like xylometazoline produce decongestion of nasal mucosa and may make insertion of bronchoscope easier. The addition of topical vasoconstrictor to lignocaine may have advantage in terms of patient comfort and for reducing local complications. Although evaluated in the settings of nasal endoscopy and nasotracheal intubation, randomized trials on the role of topical vasoconstrictors during flexible bronchoscopy are not available. The aim of this randomized trial is to study the effect of topical nasal xylometazoline administration during flexible bronchoscopy.

DETAILED DESCRIPTION:
Study design: Randomized double-blind placebo controlled study Study setting: Bronchoscopy room in Department of pulmonary medicine and sleep disorders at AIIMS, New Delhi Sample size: 200 patients (100 in each arm)

Inclusion criteria:

a) All adults > 18 years of age undergoing flexible bronchoscopy via nasal route

Exclusion criteria:

1. Uncontrolled hypertension
2. coronary artery disease

b) Pregnancy c) refusal of consent d) Hypoxemia (oxygen saturation [by pulse oximetry] < 92% with Fio2 of ≥ 0.3 e) Bronchoscopy not performed by nasal route f) Bronchoscopy performed through an artificial airway

Randomisation:

Computer generated Block randomisation with block size of 10 will be used to generate list of random numbers based on which subjects will be allocated to either of the groups.

Procedure of study The operator, assistant, drug administrator and outcomes assessor will be blinded. Patients meeting eligibility criteria will be randomized to receive either study drug Xylometazoline (0.1% nasal drops) (Otrivin, Novartis) (3 drops into each nostril) or 0.9% saline (3 drops into each nostril) placebo. This will be administered as ten minutes before bronchoscopy. This will be followed by the standard topical anesthesia procedure followed in our institution involving 5ml of 2% lignocaine gel into the nostril and 4 sprays of 10% lignocaine to the pharynx. Nebulized lignocaine shall not be administered. Transnasal flexible bronchoscopy will be performed with additional 1% lignocaine solution administered as "spray as you go" method. All diagnostic procedures or airway inspection procedures will be included. Patients shall undergo hemodynamic monitoring throughout the procedure. Procedures shall be performed without administration of upfront sedation and intraprocedural sedation shall be at the discretion of the operator.

Data will be recorded on a predesigned proforma. Baseline patient characteristics will be compared between the two groups. Categorical variables will be summarised by frequency (%) and chi-square test of proportion will be used to compare between the two groups.Quantitative variables will be summarised by mean±SD or median(IQR),as appropriate. Student's t-test or Wilcoxon rank sum test as appropriately be used to compare distribution of quantitative variables between the two groups. Stata statistical software will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

- All adults > 18 years of age undergoing flexible bronchoscopy via nasal route

Exclusion criteria:

* Uncontrolled hypertension
* coronary artery disease
* Pregnancy
* refusal of consent
* Hypoxemia (oxygen saturation [by pulse oximetry] < 92% with Fio2 of ≥ 0.3
* Bronchoscopy not performed by nasal route
* Bronchoscopy performed through an artificial airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Operator rated difficulty in nasal bronchoscope negotiation (VAS) | At study completion approximately 4 months
  Visual Analogue scale

SECONDARY OUTCOMES:
Assistant rated Faces Pain scale for discomfort on nasal bronchoscope insertion | At study completion approximately 4 months
  10 point scale divided into six categories
Patient rated nasal pain on procedure completion (VAS) | At study completion approximately 4 months
  Visual Analogue scale
Operator rated nasal mucosal trauma (VAS) | At study completion approximately 4 months
  Visual Analogue scale
Complications | At study completion approximately 4 months
  Proportion of patients developing complications

CONTACTS AND LOCATIONS:
Overall Officials: Karan Madan, MD, DM, Principal Investigator — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - AIIMS, Delhi, New Delhi
  - AIIMS, New Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sryma PB, Mittal S, Tiwari P, Mohan A, Hadda V, Guleria R, Madan K. Topical nasal xylometazoline for flexible bronchoscopy (VAIN): A randomized, double-blind, placebo-controlled trial. Respir Investig. 2021 May;59(3):350-355. doi: 10.1016/j.resinv.2020.12.004. Epub 2021 Jan 29. PMID 33518471